CLINICAL TRIAL: NCT06789120
Title: Acute Effects of Instrument-assisted Soft Tissue Mobilization on the Flexibility, Strength, Vertical Jump, and Dynamic Balance Performances of the Plantar Flexor Muscle in Professional Football Players.
Brief Title: Acute Effects of Instrument-assisted Soft Tissue Mobilization in Football Players
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Karabuk University (Other)
Collaborators: The Scientific and Technological Research Council of Turkey (Other)
Responsible Party: Principal Investigator, METEHAN YANA, Director, Karabuk University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Sport health
Record Dates: First submitted 2025-01-13; First posted 2025-01-23 (Actual); Last update posted 2025-01-23 (Actual); Status verified 2025-01

CONDITIONS: Myofascial Pain
Keywords: Myofascial release; plantar flexors; Soccer player; Balance

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Treatment Group (Experimental): In the study, the Graston device will be applied to the plantar flexor muscles of the patients. The medial and lateral gastarosoleus muscles and tendon will be applied deeply for 3 minutes, and the soleus muscle will be applied deeply for 90 seconds.
  Interventions: Other: Instrument-assisted soft tissue mobilization

INTERVENTIONS:
Other: Instrument-assisted soft tissue mobilization — In the study, the Graston device will be applied to the plantar flexor muscles of the patients. The medial and lateral gastarosoleus muscles and tendon will be applied deeply for 3 minutes, and the soleus muscle will be applied deeply for 90 seconds.

SUMMARY:
For professional footboll players, the balance, jumping, and performance capabilities of the plantar flexor muscle group are crucial on the field. Performance-enhancing interventions for these muscles are essential for improving player performance, preventing injuries, and accelerating the rehabilitation process. limitations and myofascial problems often occur in these muscles due to overuse and fatigue. Graston technique (GT), one of the instrument-assisted soft tissue mobilization techniques (IASTM), is thought to be an effective method in sports rehabilitation by accelerating relaxation and blood flow. However, this situation has not been adequately examined in the literature. Therefore, we think that the results of this study will provide an important perspective to the literature.

DETAILED DESCRIPTION:
The plantar flexors (PF) and the ankle joint are of great importance as they play an essential role in generating force on the ground. The ankle PF is the primary structure where energy is stored and released during movement and is the primary source of forward propulsion. This constitutes an important source of power for soccer players. Ankle flexibility is linked to dynamic balance capacity, which influences important elements such as speed, kick accuracy, ball control and agility. Muscle tension, myofascia and reduced range of motion (ROM) are frequently observed in team sports such as soccer, which increases the frequency of muscle injuries. Studies have shown that movement efficiency is reduced when movement is restricted in both the lower and upper limbs. Therefore, preservation and restoration of ROM is important to minimize injuries and improve performance, and myofascial release is often used in this context. Instrument-assisted soft tissue mobilization-Graston Technique (IASTM-GT) entails repetitive mechanical stimulation, including compression and shear stress applied to soft tissues such as muscles, deep fascia and tendons. It facilitates the healing process by creating microtrauma, disrupting collagen connections, increasing blood circulation and promoting cellular regeneration.Numerous studies have extensively investigated the flexibility effect of Graston Technique (GT) on athletes, particularly by improving ROM and accelerating the recovery process in key muscle groups such as the thighs, quadriceps and plantar flexors (PF). However, the evidence is not clear on how GT specifically affects the function of the PF muscle and its implications on the performance and health of football players. The effectiveness of facial mobilization in football players may be important for improving athlete performance and injury prevention. The results of this study may guide healthcare professionals by providing information about the effectiveness of these non-invasive techniques in athlete performance, treatment and rehabilitation process in clinical practice. In this context, the aim of this study was to investigate the acute effect of fascial release applied to the PF muscles on ROM, jumping ability and muscle strength.

ELIGIBILITY:
Inclusion Criteria:

* Healthy professional male football players

Exclusion Criteria:

* Having a medical history of chronic disease (cardiopulmonary, neurological, thyroid gland diseases)
* Having acute musculoskeletal system problems
* No disability or surgical intervention in the lower extremity in the last year.

Ages: 18 Years to 30 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2023-12-05 (Actual); Primary Completion 2024-03-10 (Actual); Study Completion 2024-03-10 (Actual)

PRIMARY OUTCOMES:
Range of motion | baseline, immediately after the intervention
  Dorsiflexion Reng Of Motion tests were conducted using a handheld manual goniometer.
Muscle strength | baseline, immediately after the intervention
  The handheld dynamometer (Model: Activ5-M\ Activforce2) was used to measure isometric strength in the Plantar flexors of ankle.
Balance | baseline, immediately after the intervention
  The Y Balance Test (YBT) was employed for evaluating dynamic balance across three reach directions: anterior (ANT), posteromedial (PM), and posterolateral (PL)
Jump Performance | baseline, immediately after the intervention
  My Jump 2, a mobile app designed for vertical jump performance, high-speed video capture

CONTACTS AND LOCATIONS:
Overall Officials: Metehan Yana, PhD, Study Chair — Karabuk University
Locations (2):
- Turkey (Türkiye) (2):
  - Karabük University, Karabük, Karabük Province
  - Karabük University, Karabük

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Vardiman JP, Siedlik J, Herda T, Hawkins W, Cooper M, Graham ZA, Deckert J, Gallagher P. Instrument-assisted soft tissue mobilization: effects on the properties of human plantar flexors. Int J Sports Med. 2015 Mar;36(3):197-203. doi: 10.1055/s-0034-1384543. Epub 2014 Oct 27. PMID 25347141
- [Background] Laudner K, Compton BD, McLoda TA, Walters CM. Acute effects of instrument assisted soft tissue mobilization for improving posterior shoulder range of motion in collegiate baseball players. Int J Sports Phys Ther. 2014 Feb;9(1):1-7. PMID 24567849
- [Background] Nazary-Moghadam S, Yahya-Zadeh A, Zare MA, Ali Mohammadi M, Marouzi P, Zeinalzadeh A. Comparison of utilizing modified hold-relax, muscle energy technique, and instrument-assisted soft tissue mobilization on hamstring muscle length in healthy athletes: Randomized controlled trial. J Bodyw Mov Ther. 2023 Jul;35:151-157. doi: 10.1016/j.jbmt.2023.04.079. Epub 2023 Apr 21. PMID 37330762